CLINICAL TRIAL: NCT03590496
Title: Safety and Efficacy of PROPionatE for Reduction of LDL Cholesterol (PROPER-LDL Trial) - A Phase 2 Randomized Placebo Controlled Double-blind Trial
Brief Title: Safety and Efficacy of Propionate for Reduction of LDL Cholesterol
Acronym: PROPER-LDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Arash Haghikia, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PROPER-LDL Trial
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hypercholesterolemia
Keywords: propionate
MeSH Terms: conditions — Hypercholesterolemia | interventions — Propionates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): 31 patients will be treated with 500mg Calcium-Propionate capsules (twice a day) for 8 weeks.
  Interventions: Dietary Supplement: Calcium-Propionate 500mg
- Arm 2 (Placebo Comparator): 31 patients will be treated with placebo capsules (twice a day) for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Calcium-Propionate 500mg — Calcium-Propionate capsules
  Arms: Arm 1
Other: Placebo — Placebo capsules without any active ingredient
  Arms: Arm 2

SUMMARY:
The objective of the trial is to evaluate a potential impact of food supplements with the short chain fatty acid propionate on blood LDL cholesterol level.

DETAILED DESCRIPTION:
62 patients with low cardiovascular risk will be 1:1 randomized to receive either placebo (b.i.d.) or 500mg of propionate (b.i.d.). The primary endpoint is the change (delta) in blood LDL cholesterol levels after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with hypercholestrolemia and a LDL serum level of > 115 mg/dl
* age of patient between 20 and 70 years
* participant is fully competent and has given his/her written informed consent to the scheduled trial conduct

Exclusion Criteria:

* patients with acute coronary syndrome in the last 4 weeks
* patients with chronic symptomatic heart failure (NYHA 2-4)
* patients with chronic renal failure and a GFR < 45 ml/min
* patients with chronic liver disease
* patients with hematological diseases
* patients with severe diseases of other organ systems (tumors, infections)
* pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol reduction | 8 weeks
  mg/dL

SECONDARY OUTCOMES:
total cholesterol | 8 weeks
  mg/dL
HDL-cholesterol | 8 weeks
  mg/dL
non HDL | 8 weeks
  mg/dL
Ratio HDL/LDL | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arash Haghikia, PD MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yusuf S, Bosch J, Dagenais G, Zhu J, Xavier D, Liu L, Pais P, Lopez-Jaramillo P, Leiter LA, Dans A, Avezum A, Piegas LS, Parkhomenko A, Keltai K, Keltai M, Sliwa K, Peters RJ, Held C, Chazova I, Yusoff K, Lewis BS, Jansky P, Khunti K, Toff WD, Reid CM, Varigos J, Sanchez-Vallejo G, McKelvie R, Pogue J, Jung H, Gao P, Diaz R, Lonn E; HOPE-3 Investigators. Cholesterol Lowering in Intermediate-Risk Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2021-31. doi: 10.1056/NEJMoa1600176. Epub 2016 Apr 2. PMID 27040132
- [Background] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Background] Kataoka Y, St John J, Wolski K, Uno K, Puri R, Tuzcu EM, Nissen SE, Nicholls SJ. Atheroma progression in hyporesponders to statin therapy. Arterioscler Thromb Vasc Biol. 2015 Apr;35(4):990-5. doi: 10.1161/ATVBAHA.114.304477. Epub 2015 Feb 26. PMID 25722430
- [Background] Berggren AM, Nyman EM, Lundquist I, Bjorck IM. Influence of orally and rectally administered propionate on cholesterol and glucose metabolism in obese rats. Br J Nutr. 1996 Aug;76(2):287-94. doi: 10.1079/bjn19960032. PMID 8813902
- [Background] Lu Y, Fan C, Li P, Lu Y, Chang X, Qi K. Short Chain Fatty Acids Prevent High-fat-diet-induced Obesity in Mice by Regulating G Protein-coupled Receptors and Gut Microbiota. Sci Rep. 2016 Nov 28;6:37589. doi: 10.1038/srep37589. PMID 27892486
- [Background] Chambers ES, Viardot A, Psichas A, Morrison DJ, Murphy KG, Zac-Varghese SE, MacDougall K, Preston T, Tedford C, Finlayson GS, Blundell JE, Bell JD, Thomas EL, Mt-Isa S, Ashby D, Gibson GR, Kolida S, Dhillo WS, Bloom SR, Morley W, Clegg S, Frost G. Effects of targeted delivery of propionate to the human colon on appetite regulation, body weight maintenance and adiposity in overweight adults. Gut. 2015 Nov;64(11):1744-54. doi: 10.1136/gutjnl-2014-307913. Epub 2014 Dec 10. PMID 25500202
- [Derived] Haghikia A, Zimmermann F, Schumann P, Jasina A, Roessler J, Schmidt D, Heinze P, Kaisler J, Nageswaran V, Aigner A, Ceglarek U, Cineus R, Hegazy AN, van der Vorst EPC, Doring Y, Strauch CM, Nemet I, Tremaroli V, Dwibedi C, Krankel N, Leistner DM, Heimesaat MM, Bereswill S, Rauch G, Seeland U, Soehnlein O, Muller DN, Gold R, Backhed F, Hazen SL, Haghikia A, Landmesser U. Propionate attenuates atherosclerosis by immune-dependent regulation of intestinal cholesterol metabolism. Eur Heart J. 2022 Feb 10;43(6):518-533. doi: 10.1093/eurheartj/ehab644. PMID 34597388